CLINICAL TRIAL: NCT01084642
Title: A Pilot Study Surveying Female Cancer Patients' Preference For Sexual Health Interventions
Brief Title: Female Cancer Patients' Preference For Sexual Health Interventions
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-034
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer; Gynecologic Cancer
Keywords: Survey; Sexual Health Issues; 10-034
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- survey: Participants will be asked to complete a survey as a one time assessment.

SUMMARY:
The purpose of this study is to survey female cancer patients' awareness of and preference for methods to improve sexual health. This information will help to improve our understanding of the needs and preferences for sexual health strategies and interventions of our female patients.

The findings of this survey will also be used to develop feasible sexual health resources for our patients and enhance the success of grant proposals to support future sexual health interventions at MSKCC.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to communicate in English to complete the tests.
* Study group of breast and/or gynecological cancer survivors.
* History of Primary diagnosis of breast and/or gynecological cancer
* At least 21 years of age.
* In the judgement of the consenting professional able to provide informed consent
* In the judgement of the consenting professional, able to communicate well enough in English through verbal and written communication to complete the study assessments.

Exclusion Criteria:

* In the judgement of the consenting professional, the individual is able to provide informed consent.
* Patients with a psychiatric disorder precluding response to the surveys.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinics at MSKCC
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2010-03-04 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Participant' awareness of sexual health issues & preference for sexual health intervention | 2 years

SECONDARY OUTCOMES:
To assess & describe female cancer patients' attitudes towards & preference of methods to receive sexual health information (verbal or written) & psychosexual education patient information cards or intervention modality (telephone, in-person or online). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Carter, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org